CLINICAL TRIAL: NCT03393104
Title: Effects of Patient Education and Motor Control Exercise on Selected Clinical and Psychosocial Variables Among Rural Community-dwelling Adults With Chronic Low Back Pain: a Randomized Clinical Trial
Brief Title: Patient Education and Motor Control Exercise Among Rural Community-dwelling Adults With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayero University Kano, Nigeria (Other)
Responsible Party: Principal Investigator, Aminu A. Ibrahim, Doctoral Student, Bayero University Kano, Nigeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPS/15/PPT/00009
Record Dates: First submitted 2017-12-06; First posted 2018-01-08 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Nonspecific Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Motor Control Exercise; Patient Education
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participants' treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Control Exercise and Patient Education (Experimental): Participants will receive a total of 16 sessions (2 sessions per week) of motor control exercise and 4 sessions (1 session per week) of patient education program as described in respective protocol.
  In addition, they will also perform segmental stretching exercises and instructed to perform continuous overground walk as indicated in the control group.
  Interventions: Behavioral: Motor Control Exercise; Behavioral: Patient Education
- Motor Control Exercise (Experimental): Participants will receive a total of 16 sessions (2 sessions per week) of motor control exercise aiming at improving function of specific muscles of the lumbopelvic region and the control of posture and movement.
  They will also perform segmental stretching exercises and instructed to perform continuous overground walk as indicated in the control group.
  Interventions: Behavioral: Motor Control Exercise
- Patient Education (Experimental): Participants will receive patient education session once a week at interval of 1-week over 8-weeks (4 sessions). The program will be aiming to provide non-threatening information to enable patients to better understand their pain, change any unhelpful beliefs about LBP, decrease fear avoidance behavior and catastrophic thought, promote positive attitude, self-management, and active coping strategies.
  They will also perform segmental stretching exercises and instructed to perform continuous overground walk as indicated in the control group.
  Interventions: Behavioral: Patient Education

INTERVENTIONS:
Behavioral: Motor Control Exercise — Activation of specific muscles of the lumbopelvic region responsible for providing stability or control of posture and movement.
  Other Names: Specific stabilisation exercise
  Arms: Motor Control Exercise; Motor Control Exercise and Patient Education
Behavioral: Patient Education — Education aiming to change unhelpful beliefs about LBP, decrease fear avoidance behavior and catastrophic thought, promote positive attitude, self-management, and active coping strategies.
  Other Names: Cognitive Education
  Arms: Motor Control Exercise and Patient Education; Patient Education

SUMMARY:
Low back pain (LBP) is the leading cause of years lived with disability globally with increasing concern about its impact in low- and middle-income countries like those situated in Africa where most people are living in rural areas with limited access to health care. Epidemiological studies in Nigeria suggest that the burden of chronic low back pain (CLBP) in rural areas is greater than in urban areas, with both biomechanical and psychological factors being implicated. However, despite the burden of CLBP in rural Nigeria, rehabilitation services are lacking even at the rural primary healthcare centers due to the absence of physiotherapists. Current clinical practice guidelines unanimously recommend education including instruction on self-management options, and exercise as frontline interventions to help individuals with CLBP. However, the specific content of these interventions are rarely described. Patient education (PE) strategies incorporating both biomedical and psychosocial information have been shown to be beneficial for CLBP. Moreover, exercises in the form of motor control exercises (MCEs) have been proven to be effective for CLBP. However, RCTs examining the effects of PE and MCE individually or in combination among rural community-dwelling adults with CLBP are scarce.

The purpose of this study is to determine the effects of PE and MCE program on selected clinical and psychosocial variables among rural community-dwelling adults with nonspecific CLBP.

DETAILED DESCRIPTION:
Participants will be recruited and assigned to one of three intervention groups that include PE plus MCE group, MCE group, or PE group using a block random technique based on an electronic randomization table generated by a computer software program. Blinded assessment of all outcomes will be performed at baseline, 8 weeks after randomization and at 3, 6 and 12 months follow-up.

Primary outcomes will be functional disability and pain intensity. Secondary outcomes will be quality of life, global perceived recovery, fear-avoidance beliefs, pain catastrophizing, back pain consequences beliefs, and physical performance (finger-floor test, repeated sit-to-stand test, and the 50-foot walk test) Data will be analyzed using descriptive and inferential (mixed-model ANOVA/linear mixed-effects model) statistics. All statistical analyses will be performed on IBM SPSS Statistics ver. 23.0 (IBM Co., Armonk, NY, USA) at alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female between 16 and 70 years old.
2. Primary complaint of LBP with or without leg pain experienced at least over the previous 3 months duration.
3. Mean LBP intensity at least ≥ 3 on numerical rating scale during the past week.
4. Ability to read/understand English or Hausa language.

Exclusion Criteria:

1. Previous history of thoracic spine or lumbosacral spine surgery.
2. Any neurological findings indicating radiculopathy.
3. Evidence of serious spine pathology (e.g. tumor, infection, fracture, spinal stenosis, inflammatory disease).
4. Unstable or severe disabling chronic cardiovascular and pulmonary disease.
5. History of serious psychological or psychiatric illness.
6. Current pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Change in functional disability | Baseline, 8 weeks after beginning treatment, and 3, 6 and 12 months follow-up
  Functional disability will be measured by Oswestry disability index (ODI). The questionnaire consists of 10 items with each item having six statements. All scores are summed, then multiplied by two to obtain the index (range 0 to 100) with higher score indicating greater disability.
Change in pain Intensity | Baseline, 8 weeks after beginning treatment, and 3, 6 and 12 months follow-up
  Pain Intensity will be measured by an 11-point (0-10) Numerical Pain Rating Scale (NPRS), in which 0 represents "no pain" and 10 represents "worst pain imaginable".

SECONDARY OUTCOMES:
Change in quality of life | Baseline, 8 weeks after beginning treatment, and 3, 6 and 12 months follow-up
  Quality of life will be measured using the SF-12 health survey. The questionnaire consists of 12 items questioned weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better health.
Change in global impression of recovery | Baseline, 8 weeks after beginning treatment, and 3, 6 and 12 months follow-up
  Global impression of recovery will be measured by an 11-point Global Perceived Effect Scale (GPES). it range from -5 (vastly worse) to 0 (unchanged) to +5 (completely recovered). Higher scores indicate better recovery.
Change in fear-avoidance beliefs | Baseline, 8 weeks after beginning treatment, and 3-month follow-up
  Fear avoidance beliefs will be measured by the fear-avoidance beliefs questionnaire (FABQ). The questionnaire consists of 16 self-response items, rated on a seven-point ordinal scale from 0 to 6. It also contains two subscales, a 7-item subscale concerning work, and a 4-item subscale concerning physical activity. Each subscale scores are summed giving possible ranges for the physical activity subscale of 0-24 and for the work subscale between 0-42. Higher score indicate greater fear and avoidance beliefs.
Change in pain catastrophization | Baseline, 8 weeks after beginning treatment, and 3-month follow-up
  Pain catastrophizing will be measured by the pain catastrophizing scale (PCS). The scale consists of 13 items rated on 5-point ordinal scale (0-5).The total score ranges from 0-52 with higher score indicating more catastrophic thoughts.
Change in back pain consequences beliefs | Baseline, 8 weeks after beginning treatment, and 3-month follow-up
  The back pain consequences beliefs will be measured by the Back Beliefs Questionnaire (BBQ). The BBQ is a 14-item scale, with each item rated using a 5-point Likert scale. Nine items (1, 2, 3, 6, 8, 10, 12, 13, and 14) are used for scoring of the questionnaire resulting in a total score ranging from 9-45 with lower scores indicating the more pessimistic beliefs regarding the consequences of back pain.
Change in mobility of the spine and pelvis | Baseline and 8 weeks after beginning treatment
  The finger-floor distance test (FFD) measures mobility of both the whole spine and the pelvis in the overall motion of bending forward.
Change in functional performance of sit-to-stand | Baseline and 8 weeks after beginning treatment
  The repeated sit-to-stand test measures the time taken to sit-to-stand, five times from a standard chair. The shorter the time taken to complete the test, the better the performance.
Change in functional performance of 50-foot walk | Baseline and 8 weeks after beginning treatment
  The 50-foot walk test measures time taken to walk a distance of 50-foot. The shorter the time taken to complete the test, the better the performance.

CONTACTS AND LOCATIONS:
Overall Officials: Aminu A. Ibrahim, Principal Investigator — Physiotherapy Department, Faculty of Allied Health Sciences, College of Health Sciences, Bayero University, Kano. Nigeria
Locations (1):
- Tsakuwa Primary Healthcare Center, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim AA, Akindele MO, Ganiyu SO. Effectiveness of patient education plus motor control exercise versus patient education alone versus motor control exercise alone for rural community-dwelling adults with chronic low back pain: a randomised clinical trial. BMC Musculoskelet Disord. 2023 Feb 23;24(1):142. doi: 10.1186/s12891-022-06108-9. PMID 36823567
- [Derived] Ibrahim AA, Akindele MO, Ganiyu SO, Bello B. Effects of motor control exercise and patient education program in the management of chronic low back pain among community-dwelling adults in rural Nigeria: a study protocol for a randomized clinical trial. Integr Med Res. 2019 Jun;8(2):71-81. doi: 10.1016/j.imr.2019.02.001. Epub 2019 Feb 21. PMID 31080731